CLINICAL TRIAL: NCT00421408
Title: Impact of a Protein Supplement on Bone Mass in Older Men and Women
Brief Title: The Effect of Protein Supplementation on Bone Health in Healthy Older Men and Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0610001951; R01AR053701 (NIH); 1R01AR053701-01A1 (NIH)
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Bone Resorption; Osteoporosis
Keywords: Dietary protein; Calcium; Parathyroid hormone; Bone markers; Bone mineral density; IGF-1; Urine Calcium
MeSH Terms: conditions — Bone Resorption; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protein powder (Experimental): Participants will receive a protein supplement daily (40 g whey protein supplement).
  Interventions: Dietary Supplement: Whey protein supplement
- Placebo carbohydrate (Placebo Comparator): Participants will receive a placebo supplement daily (40 g maltodextrin).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — 40-g whey protein supplement daily for 18 months
  Arms: Protein powder
Dietary Supplement: Placebo — Placebo supplement daily for 18 months
  Arms: Placebo carbohydrate

SUMMARY:
Women and men consuming a low protein diet may be at risk for bone loss. The purpose of this study is to determine whether a daily protein supplement will improve bone health among healthy older adults.

DETAILED DESCRIPTION:
Dietary protein plays an important role in maintaining balanced calcium levels in the body. Protein's impact on skeletal health remains unclear. It is well accepted that increasing dietary protein results in greater excretion of calcium through urine. The excreted calcium is thought to come in part from bone, which would suggest a negative effect on bone health. However, recent studies have found that higher protein intake is, in fact, associated with higher bone mineral density and lower rates of bone loss. The purpose of this study is to determine if a daily protein supplement will improve bone health and hormonal measures of bone metabolism among healthy older men and women who consume low-to-normal levels of dietary protein.

This study will last 18 months. For the duration of the study, participants will be randomly assigned to receive either a 40-gram protein supplement or placebo daily. There will be a total of nine study visits that will occur at screening, study entry, Month 1.5, and every three months thereafter. Dietary records, nutritional counseling, glucose finger stick tests, and questionnaires related to falls, physical activity, habits, and study satisfaction will occur at all study visits. Blood and urine collection, functional testing, and bone mineral density (BMD) testing will occur at selected visits. At Months 0 and 18, half of the participants will undergo a quantitative computed tomography (CT) scan to determine bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Willing to travel to one of the study sites
* Women age 60 years or greater, men age 70 years or greater
* Dietary protein intake level between 0.6 g/kg and 1.0 g/kg at baseline

Exclusion Criteria:

* Active Paget's disease
* Primary hyperparathyroidism or unexplained hypercalcemia
* Untreated hyperthyroidism or hyperthyroidism that has resulted from medical treatment
* Diabetes mellitus type 1
* Cancer diagnosis for solid malignancies (e.g., cancer of the colon, breast,prostate, lungs, lymphocytes) within the 18 months prior to study entry
* Long-term use of chemotherapeutic drugs, aromatase inhibitors, or tamoxifen
* Active treatment for leukemia or multiple myeloma
* Active inflammatory bowel disease
* Life expectancy of less than 2 years
* Current and ongoing use of methotrexate, phenytoin, phenobarbital, or inhaled corticosteroids at a dose of greater than 800 mcg/day
* Use of raloxifene, estrogen, androgen, progesterone, soy isoflavones, oral glucocorticoids, or herbal supplements with estrogenic activity OR a change in dosage of thyroid medications within the 1 year prior to study entry if unwilling to avoid such agents during the duration of the study
* Current use of antiresorptive agents (e.g., calcitonin or bisphosphonates). More information about this criterion can be found in the protocol.
* serum creatinine greater than 1.2 mg/dl
* History of chronic liver disease or evidence of liver disease at screening
* Bilateral hip replacement
* women who have a bone mineral density T-score < -2.5 at either the hip or spine unless they have decided to decline treatment with conventional anti-osteoporotic medications
* Body mass index (BMI) greater than 32 or less than 19
* Use of proton-pump inhibitors taken twice daily
* Fasting glucose level greater than 110 mg/dl
* Serum albumin level less than 3.0 mg/dl
* Kidney stones or history of kidney stones within the 3 years prior to study entry

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2007-02; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl L. Insogna, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale University, New Haven, Connecticut

REFERENCES:
- [Background] Newton KM, LaCroix AZ, Levy L, Li SS, Qu P, Potter JD, Lampe JW. Soy protein and bone mineral density in older men and women: a randomized trial. Maturitas. 2006 Oct 20;55(3):270-7. doi: 10.1016/j.maturitas.2006.04.011. Epub 2006 May 26. PMID 16730418
- [Background] Uenishi K, Ishida H, Toba Y, Aoe S, Itabashi A, Takada Y. Milk basic protein increases bone mineral density and improves bone metabolism in healthy young women. Osteoporos Int. 2007 Mar;18(3):385-90. doi: 10.1007/s00198-006-0228-5. Epub 2006 Oct 18. PMID 17048062
- [Derived] Kerstetter JE, Bihuniak JD, Brindisi J, Sullivan RR, Mangano KM, Larocque S, Kotler BM, Simpson CA, Cusano AM, Gaffney-Stomberg E, Kleppinger A, Reynolds J, Dziura J, Kenny AM, Insogna KL. The Effect of a Whey Protein Supplement on Bone Mass in Older Caucasian Adults. J Clin Endocrinol Metab. 2015 Jun;100(6):2214-22. doi: 10.1210/jc.2014-3792. Epub 2015 Apr 6. PMID 25844619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in June 2007 and the last participant was screened in October 2010. Subjects were recruited to the Yale Center for Clinical Investigation in New Haven, CT or the University of Connecticut Health Center in Farmington, CT.
Pre-assignment Details: Subjects were randomized 1 month after screening if they were found eligible after screening. Between screening and randomization their calcium and vitamin D intake was stabilized for baseline measurements.
Groups:
- Placebo Carbohydrate 40 g Daily for 18 Months: Participants will receive a placebo supplement daily (40 g maltodextrin).
  Placebo : Placebo supplement daily for 18 months
- Protein Powder 40 g Daily for 18 Months: Participants will receive a protein supplement daily (40 g whey protein supplement).
  Whey protein supplement : 40-g whey protein supplement daily for 18 months
Period: Overall Study
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Started | 102 | 106
Completed | 60 | 61
Not Completed | 42 | 45
Not completed — Lost to Follow-up | 30 | 20
Not completed — Discountinued from treatment/ f/u cont. | 12 | 25

BASELINE CHARACTERISTICS:
Population: Healthy older men and women with no known disorders that affect mineral metabolism and not taking drugs that alter skeletal metabolism.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months | Total
Number analyzed (Participants) | 102 | 106 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (6.4) | 69.9 (6.1) | 70.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 89 | 178
  Male | 13 | 17 | 30
Region of Enrollment [Number; unit: participants]
  United States | 102 | 106 | 208

OUTCOME MEASURES:

1. Primary Outcome: Change in Anterior-posterior Spine Bone Mass Density Measured by Dual Energy X-ray Absorptiometry (DXA) Compared to Baseline
Description: There is no absolute normative range for bone mineral density. Population norms have been established for specific races and men and women for the hip based on data collected by National Health Examination Nutrition Surveys (NHANES) and for the spine based largely on data collected by individual manufacturers. Values within 1 standard deviation of the population mean are generally considered normal. Values below 1 standard deviation from the population mean are generally considered to reflect reduced bone mass.
Time Frame: Measured at baseline and 18 months
Population: Only participants with data at the baseline and 18 month timeframe were used in the analysis.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 79 | 92
percentage change | 0.51 (0.38) | 0.51 (0.38)

2. Primary Outcome: Change in Spine Bone Mineral Density Measured by Quantitative Computed Tomography (QCT) Compared to Baseline
Description: There is no normative data for quantitative computed tomography it is based on local experience.
Time Frame: Measured at baseline and 18 months
Population: Only participants with data at the baseline and 18 month timeframe were used in the analysis. Only half of the study partipants were randomized to receive Quantitative Computed Tomography testing.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 30 | 30
percent change | -0.07 (1.08) | -2.64 (1.81)

3. Primary Outcome: Anterior-posterior Spine Bone Mineral Density Measured by Dual Energy X-ray Absorptiometry (DXA) at Baseline
Description: as for outcome 1
Time Frame: Measured at 0 months
Population: All participants were analyzed using the mixed models method.
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 102 | 106
g/cm^2 | 1.10 (0.01) | 1.13 (0.01)

4. Primary Outcome: Anterior-posterior Spine Bone Mineral Density Measured by Dual Energy X-ray Absorptiometry (DXA) at 9 Months
Description: as for outcome 1
Time Frame: Measured at 9 months
Population: All participants were analyzed using the mixed models method.
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 102 | 106
g/cm^2 | 1.14 (0.02) | 1.12 (0.01)

5. Primary Outcome: Anterior-posterior Spine Bone Mineral Density Measured by Dual Energy X-ray Absorptiometry (DXA) at 18 Months
Description: as for outcome 1
Time Frame: Measured at 18 months
Population: All participants were analyzed using the mixed models method.
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 102 | 106
g/cm^2 | 1.14 (0.02) | 1.12 (0.01)

6. Primary Outcome: Spine Bone Mineral Density Measured by Quantitative Computed Tomography (QCT) at Baseline
Description: There is no normative data for quantitative computed tomography it is based on local experience.
Time Frame: Measured at 0 months
Population: All participants were analyzed using the mixed models method. For the Quantitative Computed Tomography (QCT) test only half of the participants were randomized to receive it.
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 44 | 45
mg/cm^3 | 106 (3.72) | 103 (4.51)

7. Primary Outcome: Spine Bone Mineral Density Measured by Quantitative Computed Tomography (QCT) at 18 Months
Description: There is no normative data for quantitative computed tomography it is based on local experience.
Time Frame: Measured at 18 months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/cm^3
Arm/Group | Placebo Carbohydrate 40 g Daily for 18 Months | Protein Powder 40 g Daily for 18 Months
Number analyzed (Participants) | 44 | 45
mg/cm^3 | 106 (4.07) | 99.3 (4.29)

ADVERSE EVENTS:
Time Frame: AE data was collected from July 2007 to May 2012
Description: Gastrointestinal adverse events were assessed at times as part of a group of events.
Arm/Group | Placebo Carbohydrate Powder 40 g Daily | Protein Powder 40 g Daily
Serious Adverse Events (participants affected / at risk) | 14/102 | 4/106
Other Adverse Events (participants affected / at risk) | 46/102 | 56/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Carbohydrate Powder 40 g Daily (N=102) | Protein Powder 40 g Daily (N=106)
spinal fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
surgery for thyroid tumor (Endocrine disorders) | 1 (1) | 0 (0)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Liver cancer (Hepatobiliary disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Severe nose bleed (Vascular disorders) | 1 (1) | 0 (0)
Dramatic drop in blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Bleed (Vascular disorders) | 1 (1) | 0 (0)
Hernia surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute pancreatitits (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hip replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Carbohydrate Powder 40 g Daily (N=102) | Protein Powder 40 g Daily (N=106)
Mild to moderate gastro-intestinal upset (Gastrointestinal disorders) | 18 (18) | 31 (31)
Musculo-skeletal surgery (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Skin disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Infections (Infections and infestations) | 2 (2) | 0 (0)
Incidental findings on QCT (Investigations) | 4 (4) | 0 (0)
Diagnosed with Barret's esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decrease in glomerular filtration rate (Renal and urinary disorders) | 1 (1) | 0 (0)
Burning tongue syndrome (Investigations) | 1 (1) | 0 (0)
High blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bike accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder tumor (Renal and urinary disorders) | 1 (1) | 0 (0)
Attenuating mass in left kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Ruptured baker's cyst in knee while walking (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
restlessness (Nervous system disorders) | 1 (1) | 0 (0)
Mouth cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Difficult breathing due to atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Fluid retention (Cardiac disorders) | 0 (0) | 1 (1)
Acute renal failure following cardiac cath procedure (Renal and urinary disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 2 (2)
Elevated cholesterol (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in lower left quadrant (Gastrointestinal disorders) | 0 (0) | 1 (1)
Outpatient hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Increased duration of heart palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Dry mouth (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Basal squamous cells removed from right cheek (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bursa removed from right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruise and bleeding post blood draw (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthmatic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Broken bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitations of this study include the large attrition rate due to the length of the intervention and the difficulty in adhering to 40 grams of protein or placebo powder as a daily supplement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No